CLINICAL TRIAL: NCT03897270
Title: Photoacoustic Imaging of Human Breast
Brief Title: Photoacoustic Imaging of the Breast in Patients With Breast Cancer and Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I 60217; NCI-2019-01356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 60217 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-22; First posted 2019-04-01 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Breast Carcinoma; Healthy Subject
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (photoacoustic imaging of the breast) (Experimental): Participants undergo photoacoustic imaging of the breast over 30 minutes. At subject's discretion, imaging may repeat for a total of 10 studies, each in a separate day.
  Interventions: Procedure: Photoacoustic Imaging

INTERVENTIONS:
Procedure: Photoacoustic Imaging — Undergo photoacoustic imaging of the breast

SUMMARY:
This trial studies photoacoustic imaging of the breast in patients with breast cancer and healthy subjects. Dense breasts typically reduce the sensitivity of a mammography and also is associated with a higher risk of breast cancer. Photoacoustic tomography combines light and sound to provide more information about breast tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify photoacoustic features of breast malignancy and treatment response

OUTLINE:

Participants undergo photoacoustic imaging of the breast over 30 minutes. At subject's discretion, imaging may repeat for a total of 10 studies, each in a separate day.

ELIGIBILITY:
Inclusion Criteria:

* Women with clinically suspicious or confirmed breast cancer masses (that have not been surgically removed) and will/have already undergo/undergone breast magnetic resonance imaging (MRI).

Exclusion Criteria:

* Pregnant women (there are no known risks to these procedures, but any unforeseen risks are as yet undetermined, so pregnant women will be excluded by means of a verbal confirmation at time of screening).
* Women who have had breast implants in the previous 6 months.
* Women who have had lumpectomy
* Adults unable to consent.
* Individuals who are not yet adults (infants, children, teenagers).
* Pregnant women.
* Prisoners.
* There is no direct benefit of the study to any subject either non-English or English speaker. To facilitate the consent process, we will exclude non-English speaking subjects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Identify photoacoustic features of breast malignancies | Up to 3 years
  Photoacoustic excitation and detection will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Ermelinda Bonaccio, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States